CLINICAL TRIAL: NCT04895592
Title: Preoperative Radiosurgery for Brain Metastases Planned for Surgical Resection: a Two Arm Pilot Study
Brief Title: Radiosurgery Before Surgery for the Treatment of Brain Metastases
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Zachary Buchwald, Principal Investigator, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001896; NCI-2021-02761 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00001896; RAD5234-21 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2021-05-17; First posted 2021-05-20 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Metastatic Malignant Neoplasm in the Brain; Metastatic Malignant Solid Neoplasm
MeSH Terms: conditions — Brain Neoplasms; Neoplasm Metastasis | interventions — Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (SRS, low dose dexamethasone, surgery) (Experimental): Patients undergo SRS to the brain metastasis for 1-3 fractions over 1-5 days. Patients also receive low dose dexamethasone PO or IV for 2-21 days until the day of surgical resection. Patients then undergo surgical resection.
  Interventions: Drug: Dexamethasone; Procedure: Resection; Radiation: Stereotactic Radiosurgery
- Arm B (SRS, high dose dexamethasone, surgery) (Experimental): Patients undergo SRS to the brain metastasis for 1-3 fractions over 1-5 days. Patients also receive high dose dexamethasone PO or IV for 2-21 days until the day of surgical resection. Patients then undergo surgical resection.
  Interventions: Procedure: Resection; Radiation: Stereotactic Radiosurgery

INTERVENTIONS:
Drug: Dexamethasone — Given PO or IV
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
  Arms: Arm A (SRS, low dose dexamethasone, surgery)
Procedure: Resection — Undergo surgical resection
  Other Names: Surgical Resection
Radiation: Stereotactic Radiosurgery — Undergo SRS
  Other Names: Stereotactic External Beam Irradiation; stereotactic external-beam radiation therapy; Stereotactic Radiation Therapy; Stereotactic Radiotherapy; stereotaxic radiation therapy; stereotaxic radiosurgery

SUMMARY:
This early phase I trial identifies the side effects of stereotactic radiosurgery before surgery in treating patients with cancer that has spread to the brain (brain metastases). Radiation may stimulate an anti-tumor immune response. Giving stereotactic radiosurgery before surgery may reduce the risk of the cancer coming back after surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the safety of pre-operative stereotactic radiosurgery (SRS) followed by surgery for brain metastasis.

SECONDARY OBJECTIVES:

I. To evaluate the immune niche in brain metastasis following SRS in the presence of low or high dose dexamethasone.

II. To evaluate the impact of pre-operative SRS on survival outcomes.

OUTLINE: Patients are assigned to 1 of 2 arms.

ARM A: Patients undergo SRS to the brain metastasis for 1-3 fractions over 1-5 days. Patients also receive low dose dexamethasone orally (PO) or intravenously (IV) for 2-21 days until the day of surgical resection. Patients then undergo surgical resection.

ARM B: Patients undergo SRS to the brain metastasis for 1-3 fractions over 1-5 days. Patients also receive high dose dexamethasone PO or IV for 2-21 days until the day of surgical resection. Patients then undergo surgical resection.

After completion of study intervention, patients are followed up for 120 days, and then every 12 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Prior or suspected diagnosis of malignancy
* Brain metastases visible on contrasted magnetic resonance imaging (MRI) brain
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Life expectancy > 12 weeks as determined by the investigator
* Patients must have adequate organ function as determined by Neurosurgery to undergo surgery
* Willingness and ability of the subject to comply with scheduled visits, study procedures, and study restrictions
* Evidence of a personally signed informed consent indicating that the subject is aware of the neoplastic nature of the disease and has been informed of the procedures to be followed, the experimental nature of the therapy, alternatives, potential risks and discomforts, potential benefits, and other pertinent aspects of study participation
* Patient must have a negative pregnancy test, be actively taking oral contraceptives or have undergone a hysterectomy

Exclusion Criteria:

* Patients on any immunosuppressive medication other than dexamethasone
* Patients who are receiving any other investigational agents or an investigational device within 21 days before administration of first dose of study drugs
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Human immunodeficiency virus (HIV)-positive
* Pregnant or nursing women are excluded
* Prior whole brain radiotherapy or SRS to the same site planned for surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-07-20 (Actual); Primary Completion 2026-02-19 (Estimated); Study Completion 2027-02-19 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events grade 3 or greater | At 4 months post-treatment
  Evaluated using Common Terminology Criteria for Adverse Events. Tolerability of this regimen will be defined as < 33% of patients develop grade > 3 at 4 months. Adverse events will be summarized descriptively using frequencies and percentages.

SECONDARY OUTCOMES:
Density of immune niche in brain metastases | Up to 2 years
  Niche density will be assessed by immunofluorescence as described above. It will be summarized descriptively as the percent of tumor occupied by immune niche for each treatment arm, and will be compared between Arms A and B using a two-sample t-test or non-parametric equivalent, such as Mann-Whitney U test.
Time to local recurrence (LR) | From pre-operative stereotactic radiosurgery (SRS) to intracranial progression at the treated site, assessed up to 2 years
  LR will be estimated using the Kaplan-Meier method, and a 95% confidence interval for median LR will be estimated using the Brookmeyer-Crowley approach.
Time to anywhere brain failure (ABF) | From preoperative SRS to intracranial progression at any site within the brain, assessed up to 2 years
  ABF will be estimated using the Kaplan-Meier method, and a 95% confidence interval for median TBF will be estimated using the Brookmeyer-Crowley approach.
Overall survival (OS) | From pre-operative SRS initiation to death, assessed up to 2 years
  OS will be estimated using the Kaplan-Meier method, and a 95% confidence interval for median OS will be estimated using the Brookmeyer-Crowley approach.

CONTACTS AND LOCATIONS:
Overall Officials: Zachary Buchwald, MD, PhD, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (1):
- Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Jansen CS, Pagadala MS, Cardenas MA, Prabhu RS, Goyal S, Zhou C, Chappa P, Vo BT, Ye C, Hopkins B, Zhong J, Klie A, Daniels T, Admassu M, Green I, Pfister NT, Neill SG, Switchenko JM, Prokhnevska N, Hoang KB, Torres MA, Logan S, Olson JJ, Nduom EK, Del Balzo L, Patel K, Burri SH, Asher AL, Wilkinson S, Lake R, Kesarwala AH, Higgins KA, Patel P, Dhere V, Sowalsky AG, Carter H, Khan MK, Kissick H, Buchwald ZS. Pre-operative stereotactic radiosurgery and peri-operative dexamethasone for resectable brain metastases: a two-arm pilot study evaluating clinical outcomes and immunological correlates. Nat Commun. 2024 Oct 14;15(1):8854. doi: 10.1038/s41467-024-53034-6. PMID 39402027